CLINICAL TRIAL: NCT02266472
Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Metformin Extended Release (10 mg/1000 mg) Compared With the Free Combination of Empagliflozin and Metformin Extended Release Tablets in Healthy Subjects Following a High-fat, High-caloric Meal (an Open-label, Randomised, Single Dose, Crossover Trial)
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Metformin Extended Release Compared With Mono Compound Tablets in Healthy Male and Female
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.28; 2014-002360-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; empagliflozin

ARMS (2):
- Fixed dose combination (Experimental): Single dose empagliflozin/metformin
  Interventions: Drug: empagliflozin/metformin
- Single tablets combination (Active Comparator): single doses empagliflozin and metformin
  Interventions: Drug: metformin; Drug: empagliflozin

INTERVENTIONS:
Drug: metformin — single dose of metformin given as tablets
  Arms: Single tablets combination
Drug: empagliflozin/metformin — Single dose empagliflozin/metformin given as fixed-dose combination tablet
  Arms: Fixed dose combination
Drug: empagliflozin — single dose of empagliflozin given as tablet
  Arms: Single tablets combination

SUMMARY:
The purpose of this trial is to investigate bioequivalence of a newly developed fixed dose combination (FDC) tablet containing empagliflozin and metformin extended release compared to the free combination of empagliflozin and metformin extended release under fed conditions.

ELIGIBILITY:
Inclusion criteria:

* Healthy male and female subjects
* age of 18 to 55 years
* body mass index (BMI) of 18.5 to 29.9 kg/m2
* additional inclusion criteria may apply

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg or diastolic blood pressure outside the range of 50 to 90 mmHg or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (including but not limited to any kind of seizures and stroke), and other relevant neurological disorders or psychiatric disorders
* additional exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, randomised, 2-way crossover trial with 2 treatments (T and R) and 2 treatment sequences (T_R and R_T). Trial drug administrations of the 2 single dose treatments were separated by a washout period of at least 7 days.
Groups:
- Fed 10mg+1000mg Fixed Dose Combination (FDC)/Single (TR): Subjects received in period 1 a single dose of 10 mg empagliflozin/1000 mg metformin hydrochloride (HCl) extended release (XR) (1 tablet) with 240 mL of water after intake of a high-fat, high-caloric meal, followed in period 2 with a single dose of 10 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal. 2 treatments separated by a wash-out period of at least 7 days.
- Fed 10mg+1000mg Single/FDC (RT): Subjects received in period 1 a single dose of 10 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal, followed in period 2 with a single dose of 10 mg empagliflozin/1000 mg metformin HCl XR (1 tablet) with 240 mL of water after intake of a high-fat, high-caloric meal. 2 treatments separated by a wash-out period of at least 7 days.
Period: Period 1+ Washout
Arm/Group | Fed 10mg+1000mg Fixed Dose Combination (FDC)/Single (TR) | Fed 10mg+1000mg Single/FDC (RT)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2+ Washout
Arm/Group | Fed 10mg+1000mg Fixed Dose Combination (FDC)/Single (TR) | Fed 10mg+1000mg Single/FDC (RT)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS was made up of all randomised subjects who were documented to have received the trial medication.
Groups:
- Fed 10mg+1000mg FDC/Single (TR): Subjects received in period 1 a single dose of 10 mg empagliflozin/1000 mg metformin hydrochloride (HCl) extended release (XR) (1 tablet) with 240 mL of water after intake of a high-fat, high-caloric meal, followed in period 2 with a single dose of 10 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal. 2 treatments separated by a wash-out period of at least 7 days.
- Total: Total of all reporting groups
Arm/Group | Fed 10mg+1000mg FDC/Single (TR) | Fed 10mg+1000mg Single/FDC (RT) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (8.1) | 33.7 (10.1) | 33.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz of Empagliflozin in Plasma
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz)
Time Frame: -1:00 hour(h) before the drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 4:00h, 5:00h, 6:00h, 7:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h and 72:00h after drug administration
Population: Pharmacokinetic set (PKS) included all treated subjects that provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of the pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Fed 10mg+ 1000mg FDC (T): Subjects received a single dose of 10 mg empagliflozin/1000 mg metformin HCl XR (1 tablet) with 240 mL of water after intake of a high-fat, high-caloric meal.
- Fed 10mg+1000mg Single (R): Subjects received a single dose of 10 mg empagliflozin (1 tablet) together with a single dose of 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal.
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 30 | 30
nmol*h/L | 2190 (18.1) | 2210 (16.3)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based on 2-sided 90% CIs for the ratios (test to reference treatment) of the adjusted gMeans of the primary endpoints, with acceptance range of 80.00 to 125.00 %; p < 0.0001, ANOVA; ANOVA model on the logarithmic scale including random effects for 'subjects within sequences' & fixed effect for 'sequence', 'period' & 'treatment'; ratio of the adjusted means = 99.11, 90% CI 2-sided [96.40 to 101.89], Standard Deviation 6.3 — Relative bioavailability of empagliflozin was estimated by the adjusted gMean ratio of Fed 10mg+1000mg FDC divided by Fed 10mg+1000mg Single. Standard deviation is actually intraindividual geometric coefficient variation (gCV)

2. Primary Outcome: AUC0-tz of Metformin in Plasma
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 29 | 30
ng*h/mL | 10800 (20.1) | 10700 (22.4)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based on 2-sided 90% confidence intervals (CIs) for the ratios (test to reference treatment) of the adjusted geometric means (gMeans) of the primary endpoints,using an acceptance range of 80.00 to 125.00 %; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the adjusted means = 101.25, 90% CI 2-sided [96.54 to 106.19], Standard Deviation 10.7 — Relative bioavailability of metformin was estimated by the adjusted gMean ratio of Fed 10mg+1000mg FDC divided by Fed 10mg+1000mg Single. Standard deviation is actually intraindividual geometric coefficient variation (gCV)

3. Primary Outcome: Cmax of Empagliflozin in Plasma
Description: Maximum measured concentration of the empagliflozin in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 30 | 30
nmol/L | 243 (23.1) | 245 (20.4)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based on 2-sided 90% CIs for the ratios (test to reference treatment) of the adjusted gMeans of the primary endpoints, with acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the adjusted means = 99.12, 90% CI 2-sided [93.69 to 104.87], Standard Deviation 12.9 — Relative bioavailability of empagliflozin was estimated by the adjusted gMean ratio of Fed10mg+1000mg FDC divided by Fed10mg+1000mg Single. Standard deviation is actually intraindividual geometric coefficient variation (gCV)

4. Primary Outcome: Cmax of Metformin in Plasma
Description: Maximum measured concentration of the metformin in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 29 | 30
ng/mL | 1170 (25.5) | 1080 (25.2)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the adjusted means = 108.58, 90% CI 2-sided [104.17 to 113.17], Standard Deviation 9.3 — Relative bioavailability of metformin was estimated by the adjusted gMean ratio of Fed10mg+1000mg FDC divided by Fed10mg+1000mg Single. Standard deviation is actually intraindividual geometric coefficient variation (gCV)

5. Secondary Outcome: AUC0-infinity of Empagliflozin in Plasma
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 30 | 30
nmol*h/L | 2230 (18.0) | 2260 (16.3)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the adjusted means = 98.89, 90% CI 2-sided [96.18 to 101.67], Standard Deviation 6.3 — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: AUC0-infinity of Metformin in Plasma
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fed 10mg+ 1000mg FDC (T) | Fed 10mg+1000mg Single (R)
Number analyzed (Participants) | 29 | 30
ng*h/mL | 11000 (20.8) | 10800 (22.7)
Statistical Analysis 1: Comparison: Fed 10mg+ 1000mg FDC (T) vs Fed 10mg+1000mg Single (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the adjusted means = 101.37, 90% CI 2-sided [96.53 to 106.45], Standard Deviation 11.0 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until the end-of-trial examination (Up to 14 days)
Arm/Group | Fed 10mg+1000mg Single (R) | Fed 10mg+ 1000mg FDC (T)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fed 10mg+1000mg Single (R) (N=30) | Fed 10mg+ 1000mg FDC (T) (N=30)
Headache (Nervous system disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes